CLINICAL TRIAL: NCT02853513
Title: Definition of a Probabilistic Model of the Evolution of an Acute Stress Disorder (ASD ) to a Posttraumatic Stress Disorder (PTSD): an Analytical Prospective Cohort Study of Patients Directly Involved in Attacks Terrorists of 13 November 2015
Brief Title: Probabilistic Risk Modeling for Disorder Post Traumatic Stress (PTSD) After the Attacks in Paris In November 2015
Acronym: BV13
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Tours (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); University of Lorraine (Other)
Responsible Party: Principal Investigator, WISSAM EL HAGE, Professor, University Hospital, Tours
Other Study IDs: 2016-A00162-49; SC16-WEH/BV13 (Registry Identifier: Ref study CPP)
Record Dates: First submitted 2016-07-03; First posted 2016-08-03 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The scientific approach of this project proposes to build a cohort of "psychological injuries" post-attack of 13 November 2015. This is called patients "involved", ie patients who directly witnessed the events and having the most either came under automatic gunfire or were close to an explosion, whether or not physically injured.

The main objective is to define and validate a model of transition from acute stress disorder (ASD) to posttraumatic stress disorder (PTSD) for better detection of the risk of unfavorable and thus better patient supported.

The first step is to determine independent risk factors found in analytic prospective cohort study.

Bayesian models are well suited to exercise because they can integrate (i) the context related to the patient, (ii) the context related to the trauma itself, and (iii) the immediate reactions and long-term to the latter . They are particularly suited to understanding the brain disordered by saying down information (prior probability) wrong by improper memory of the traumatic event. The confrontation of these descending information and perceived bottom-information could be partly responsible for the symptoms of PTSD.

Once validated, the model will characterize the individual level the most at risk of unfavorable patients (calculating a probability of developing PTSD) and to assess the epidemiological impact on long-term cohort of event considered.

These determinations are necessary prerequisites to optimize the means of support for these current and future casualties.

The investigators main objective is to define a Bayesian model describing a resilient functioning facing a trauma which also allows to describe a possible evolution of the ASD to PTSD by an error.

The state of PTSD or not will be determined by the PCL-S scale.

DETAILED DESCRIPTION:
cohort tracking study

ELIGIBILITY:
Inclusion Criteria:

* patients who directly witnessed the events and having the most either came under automatic gunfire or were close to an explosion, whether or not physically injured

Exclusion Criteria:

* persons not physically present on the premises at the time of the attacks.
* Inability to understand or read French.
* Persons unable to express personal consent under whose major legal or private protection of liberty by judicial or administrative decision , or hospital emergency or without their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a cohort of "psychological injuries" post-attack of 13 November 2015. This is called patients "involved", ie patients who directly witnessed the events and having the most either came under automatic gunfire or were close to an explosion, whether or not physically injured.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Post traumatic disorder check list | 6 months after trauma
  PTSD diagnose

SECONDARY OUTCOMES:
Hamilton depression scale | 6 months after trauma
  personality

IPD SHARING:
Plan to Share IPD: Undecided